CLINICAL TRIAL: NCT06865560
Title: Emotional Awareness and Expression Therapy for Chronic Pain and Opioid Use Disorder - A Pilot Study
Brief Title: Emotional Awareness and Expression Therapy for Chronic Pain and Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Sturgeon, Clinical Assistant Professor of Anesthesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00266504
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Opioid Use Disorder
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional Awareness and Expression Therapy (EAET) (Experimental): Adults with chronic pain and mild to moderate opioid use disorder (OUD).
  Interventions: Behavioral: Emotional Awareness and Expression Therapy (EAET)

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy (EAET) — A validated, 8-week, group-based telehealth-based behavioral intervention for chronic pain. Session content will include pain neuroscience education, emotion-focused expressive writing, in-vivo emotional expression practices, self-compassion and forgiveness exercises, and assertive communication strategies. Participants will also be provided handouts and pre-recorded guided imagery and cognitive exercises that they can use to facilitate between-session practices.

SUMMARY:
The study is intended to test whether a group-based Zoom behavioral treatment can help adults with chronic pain and opioid use disorder (OUD) learn effective strategies for reducing pain, disability and other problems that can come with these conditions (such as depression, anxiety, and difficulty managing emotions).

DETAILED DESCRIPTION:
Emotional Awareness and Expression Therapy (EAET) is a behavioral therapy that focuses on reducing chronic pain by helping people work on the effects of stress, trauma, and emotions that they have experienced in their lives. It is delivered in group sessions of 5-7 individuals by trained therapists who treat emotions or problems in relationships to reduce chronic pain. Pain decreases through increased recognition and expression of emotions, and learning to feel safe in the presence of emotions.

The primary aim of the study is to demonstrate the feasibility, acceptability, and preliminary efficacy of the proposed EAET intervention in adults with chronic pain and opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read, write and speak English
* Have Internet access and audio-visual conferencing capability (e.g., Zoom meetings by phone or computer) in the home
* Widespread pain and has opioid use disorder (OUD)

Exclusion Criteria:

* Diagnosis of autoimmune disease, spinal cord injury, cancer.
* Currently receiving cognitive-behavioral therapy, EAET, or other psychological therapies for pain
* Open litigation regarding chronic pain in the past 1 year, as assessed in preliminary study screening.
* Inability to provide informed consent and complete study procedures (e.g., indications of suspected major cognitive impairment via observations of study staff during consenting) that would preclude comprehension or participation in study protocols.
* Pregnant or breastfeeding
* Any other diseases or conditions that would make a patient unsuitable for study participation as determined by the site principal investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Mean scores on the Treatment Acceptability and Adherence Scale (TAAS) at the post intervention timepoint. | Approximately day 70
  The TAAS is a validated instrument for behavioral interventions. Although no validated cutoff scores exist for this measure, prior research has used an informal cutoff score at the midpoint of the total score (i.e., 35 out of a possible 70) as a measure of moderate acceptability. If the EAET intervention is ineffective, low acceptability may be an explanatory factor. - scores above the midpoint - 35 out of 70 - will denote moderate acceptability of the intervention
Feasibility: Session attendance | Approximately day 70
Feasibility: Combined completion of in-session and between-session practices | Approximately day 70

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI) pain intensity | Day 1 and up to day 160
  The BPI pain intensity is a validated 4-item measure of pain intensity.
  Change is measured from day 1 to day 70 AND day 1 to day 160
Change in Pain-related OUD Exacerbation Scale (PrOUD-ES) | Day 1 and up to day 160
  Validated 4-item scale assessing self-reported degree of pain-related OUD symptom exacerbation.
  Change is measured from day 1 to day 70 AND day 1 to day 160
Change in Opioid Craving Visual Analog Scale (OC-VAS) | Day 1 and up to day 160
  The OC-VAS is a validated single-item assessment utilizing 0-100 scale reflecting degree of opioid craving.
  Change is measured from day 1 to day 70 AND day 1 to day 160
Change in Current Opioid Misuse Measure-Brief (COMM-9) | Day 1 and up to day 160
  The Comm-9 is a validated 9-item self-report measure of opioid misuse.
  Change is measured from day 1 to day 70 AND day 1 to day 160

CONTACTS AND LOCATIONS:
Overall Officials: John Sturgeon, PhD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No